CLINICAL TRIAL: NCT01052233
Title: Effect of Arthroscopic Partial Resection of Degenerative Meniscus Tear on Development of Knee Osteoarthritis: Which is the Chicken and the Egg?
Brief Title: Development of Knee Osteoarthritis After Arthroscopic Partial Resection of Degenerative Meniscus Tear
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tampere University (Other)
Collaborators: Helsinki University Central Hospital (Other); Turku University Hospital (Other Government); Kuopio University Hospital (Other); Central Finland Hospital District (Other)
Responsible Party: Principal Investigator, Teppo Jarvinen, Principal Investigator, Tampere University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 9037/403/2006
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Osteoarthritis of the Knee; Arthroscopy; Meniscal Tear
Keywords: Sham-surgery; Development of osteoarthritis; Randomized, double-blinded, placebo-controlled
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroscopy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arthroscopic partial meniscectomy (Active Comparator): Arthroscopic partial resection of degenerative tear of medial meniscus
  Interventions: Procedure: Arthroscopic partial meniscectomy
- Arthroscopy (diagnostic) (Sham Comparator): Diagnostic arthroscopy of the knee
  Interventions: Procedure: Arthroscopy (diagnostic)

INTERVENTIONS:
Procedure: Arthroscopic partial meniscectomy — Arthroscopic partial meniscectomy of the degenerative tear of medial meniscus
  Arms: Arthroscopic partial meniscectomy
Procedure: Arthroscopy (diagnostic) — Diagnostic arthroscopy of the knee
  Arms: Arthroscopy (diagnostic)

SUMMARY:
It has been previously demonstrated that the risk for the development of knee osteoarthritis is increased after both meniscus tear and meniscectomy. However, it is still unclear whether this is due to the meniscus tear per se, the surgery, or whether the development of knee osteoarthritis is completely independent of the two. Accordingly, the aim of the study is to investigate the effect of arthroscopic partial meniscectomy on the development of knee osteoarthritis 2 to 10 years after the procedure.

DETAILED DESCRIPTION:
It has been previously demonstrated that the risk for the development/progression of knee osteoarthritis is increased after both meniscus tear and meniscectomy. However, it is still unclear whether this is due to the meniscus tear per se (i.e., adverse mechanical effect on knee cartilage), the surgery (resection of the meniscus, and subsequent loss of cushion within the knee), or whether the development of knee osteoarthritis is completely independent of the two.

Accordingly, the aim of the study is to investigate the effect of Arthroscopic partial meniscectomy on the development of knee osteoarthritis 2 to 10 years after the procedure.

Patients included in the study will be randomized into one of two groups: arthroscopic partial meniscectomy and diagnostic arthroscopy (sham-surgery). The presence of knee osteoarthritis will be assessed preoperatively and 2, 5, and 10 years after the operation.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 35 to 65 years of age.
2. A pain located on the medial joint line of the knee that has persistent at least for 3 months.
3. Pain that can be provoked by palpation or compression of the joint line or a positive McMurray sign.
4. Tear of the medial meniscus on MRI.
5. Degenerative rupture of the medial meniscus confirmed at arthroscopy.

Exclusion Criteria:

1. Acute, trauma-induced onset of symptoms.
2. Locking or painful snapping of the knee joint.
3. A surgical operation performed on the affected knee.
4. Osteoarthritis of the medial compartment of the knee (determined by clinical criteria of the ACR).
5. Osteoarthritis on knee radiographs (Kellgren-Lawrence > 1).
6. Acute (within the previous year) fractures of the knee.
7. Decreased range of motion of the knee.
8. Instability of the knee.
9. MRI assessment showing a tumor or any other complaint requiring surgical or other means of treatment.
10. Arthroscopic assessment showing anything other than a degenerative tear of the medial meniscus requiring surgical intervention.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2010-01; Primary Completion 2016-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Radiological assessment of OA of the knee (Kellgren-Lawrence -classification) | 2 and 10 years postoperatively

SECONDARY OUTCOMES:
ACR (The American College of Rheumatology) clinical criteria for Osteoarthritis of the knee | 2 and 10 years postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Raine Sihvonen, MD, Study Chair — Tampere City Hospital; Teppo Järvinen, MD, PhD, Principal Investigator — Tampere University
Locations (5):
- Finland (5):
  - Helsinki Central Hospital, Helsinki
  - Central Finland Hospital District, Jyväskylä
  - Kuopio University Hospital, Kuopio
  - Tampere City Hospital, Tampere
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Sillanpaa N, Iivanainen M, Turkiewicz A, Sihvonen R, Paavola M, Taimela S, Jarvinen TLN, Englund M. Effect of arthroscopic partial meniscectomy on structural degeneration of the knee - A 5-year MRI-based follow-up of the placebo-surgery controlled FIDELITY (Finnish Degenerative Meniscus Lesion Study) trial. Osteoarthritis Cartilage. 2025 Feb;33(2):276-282. doi: 10.1016/j.joca.2024.09.003. Epub 2024 Sep 12. PMID 39277028
- [Derived] Sihvonen R, Paavola M, Malmivaara A, Itala A, Joukainen A, Kalske J, Nurmi H, Kumm J, Sillanpaa N, Kiekara T, Turkiewicz A, Toivonen P, Englund M, Taimela S, Jarvinen TLN; FIDELITY (Finnish Degenerative Meniscus Lesion Study) Investigators. Arthroscopic partial meniscectomy for a degenerative meniscus tear: a 5 year follow-up of the placebo-surgery controlled FIDELITY (Finnish Degenerative Meniscus Lesion Study) trial. Br J Sports Med. 2020 Nov;54(22):1332-1339. doi: 10.1136/bjsports-2020-102813. Epub 2020 Aug 27. PMID 32855201
- [Derived] Sihvonen R, Kalske R, Englund M, Turkiewicz A, Toivonen P, Taimela S, Jarvinen TLN; Finnish Degenerative Meniscal Lesion Study (FIDELITY) Investigators. Statistical analysis plan for the 5-year and 10-year follow-up assessments of the FIDELITY trial. Trials. 2020 Jan 14;21(1):76. doi: 10.1186/s13063-019-3833-2. PMID 31937344